CLINICAL TRIAL: NCT01623687
Title: Bone Forming at Prosthetic Surfaces. A Randomized Clinical F-PET/CT Study
Brief Title: Bone Forming at Prosthetic Surfaces. Fingerprint2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUllmark Apr -12
Record Dates: First submitted 2012-01-17; First posted 2012-06-20 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Osteo Arthritis
Keywords: total hip arthroplasty; bone metabolism; mineralisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regenerex (Active Comparator)
  Interventions: Device: Component for acetabulum (Regenerex RingLoc cup)
- Lub cup (Active Comparator)
  Interventions: Device: Components for the acetabulum (Lubinus cross linked cup)
- SP II (Active Comparator)
  Interventions: Device: Arthroplasty components are for the femur (Cemented Lubinus SP II stem)
- Corail (Active Comparator)
  Interventions: Device: Arthroplasty components are for the femur (Corail stem)

INTERVENTIONS:
Device: Component for acetabulum (Regenerex RingLoc cup) — A fibrous metal uncemented Regenerex RingLoc cup (Biomet, Warsaw, Il, USA)
  Other Names: Regenerex RingLoc cup
  Arms: Regenerex
Device: Components for the acetabulum (Lubinus cross linked cup) — cemented Lubinus cross linked cup (Waldemar Link, Hamburg, Germany).
  Other Names: Lubinus cross linked cup
  Arms: Lub cup
Device: Arthroplasty components are for the femur (Cemented Lubinus SP II stem) — Cemented Lubinus SP II stem (Waldemar Link, Hamburg, Germany) with a ceramic 32 mm head.
  Other Names: Cemented Lubinus SP II stem
  Arms: SP II
Device: Arthroplasty components are for the femur (Corail stem) — Uncemented HA-coated Corail stem with a ceramic 32 mm head (DePuy, Johnsson & Johnsson, USA).
  Other Names: Uncemented HA-coated Corail stem with a ceramic 32 mm head
  Arms: Corail

SUMMARY:
What is the intensity of F-PET uptake in healthy and osteo arthritic femur and acetabulum, compared to the uptake adjacent to four analyzed endoprosthetic components 1½ and 6 months after surgery?

DETAILED DESCRIPTION:
A clinical study of 26 patients, age 50-69 years, healthy unless osteoarthritis in one hip, randomized in four groups plus a reference group of same 26 patient´s contralateral healthy hip.

Intervention will be surgery with a total hip arthroplasty. The studied endoprosthetic components are: Cemented Lubinus SP II stem with a ceramic 32 mm head, a cemented Lubinus cross linked cup (Waldemar Link, Hamburg, Germany). Palacose cement with gentamycin, applied with 3:rd generation cementation technique will be used for those cemented implants.

Uncemented HA-coated Corail stem with a ceramic 32 mm head (DePuy, Johnson & Johnson, USA), a fibrous metal Regenerex RingLoc cup (Biomet, Warsaw, Il, USA) All cups will have cross linked Ultra-high-molecular-weight polyethylene (UHWMP).

Clinical score, radiography and PET uptake of Fluoride tracer (SUV) adjacent to the prosthetic surfaces will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed to have unilateral hip osteo arthritis (Charnley group A) aimed for THA at the orthopedic clinic Gävle hospital.

Exclusion Criteria:

* Systemic disease or medication affecting the skeleton

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-09 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
FEMUR: to analyze difference in SUV of the 4 upper ROI's (No 1, 7, 8 and 13) analyzed together between the cemented and uncemented groups AND: to analyze SUV of the 4 upper ROI's analyzed together between each femur study group and the reference group | 6 weeks after surgery
  There are two study groups for femur: cemented and uncemented femur prosthetic components. There are also a femur reference group.
ACETABULUM: to analyze difference in SUV of all 9 ROI's analyzed together between the cemented and uncemented acetabular study groups, and to analyze SUV of all 9 ROI's analyzed together between each acetabulum study group and the reference group | 6 weeks after surgery
  There are two study groups for acetabulum: cemented and uncemented acetabular prosthetic components. There are also an acetabular reference group.

SECONDARY OUTCOMES:
FEMUR:to analyze difference in SUV for each individual ROI inbetween the cemented and uncemented femur group | 6 weeks and 6 months
FEMUR: to analyze difference in SUV for each individual ROI between the cemented study group and the reference group. To analyze difference in SUV for each individual ROI between the uncemented study group and the reference group. | 6 weks and 6 months
FEMUR:to analyze difference in SUV for each individual ROI between the 3 time points for the cemented group. To analyze difference in SUV for each individual ROI between the 3 time points for the uncemented group. | preoperatively, 6 weeks and 6 months
FEMUR:to analyze difference in SUV for the 4 upper ROI's (No 1, 7, 8 and 13)analyzed together between the 2 study groups | 6 months
FEMUR:to analyze difference in SUV for the 4 upper ROI's analyzed together between each study group and the reference group | 6 months
ACETABULUM: to analyze difference in SUV for each individual ROI between the 2 study groups | 6 weeks and 6 months
ACETABULUM: to analyze difference in SUV for each individual ROI between the cemented study group and the reference group. To analyze difference in SUV for each individual ROI between the uncemented study group and the reference group. | 6 weeks and 6 months
ACETABULUM: to analyze difference in SUV for each individual ROI for the cemented study group between the 3 time points. To analyze difference in SUV for each individual ROI for the uncemented study group between the 3 time points. | preoperatively, 6 weeks and 6 months
ACETABULUM: to analyze difference in SUV of all 9 ROI's analyzed together between the cemented and uncemented acetabular study groups | 6 months
ACETABULUM: to analyze difference in SUV of all 9 ROI's analyzed together between the cemented and uncemented acetabular study groups, and to analyze SUV of all 9 ROI's analyzed together between each acetabulum study group and the reference group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gösta Ullmark, Study Chair — Ass Professor
Locations (1):
- Centre for research and development Uppsala university/County council of Gävleborg, Gävle, Sweden

REFERENCES:
- [Derived] Ullmark G, Sorensen J, Nilsson O, Maripuu E. Bone mineralisation adjacent to cemented and uncemented acetabular cups: analysis by [18F]-fluoride-PET in a randomised clinical trial. Hip Int. 2020 Nov;30(6):745-751. doi: 10.1177/1120700019861274. Epub 2020 Jul 19. PMID 32686502
- [Derived] Ullmark G, Sorensen J, Maripuu E, Nilsson O. Fingerprint pattern of bone mineralisation on cemented and uncemented femoral stems: analysis by [18F]-fluoride-PET in a randomised clinical trial. Hip Int. 2019 Nov;29(6):609-617. doi: 10.1177/1120700018815404. Epub 2018 Dec 6. PMID 30520317